CLINICAL TRIAL: NCT02670343
Title: Evaluation of Blood Collection Methodology Following Administration of a Single-Dose of an Oral Testosterone Undecanoate Formulation In Hypogonadal Men
Brief Title: Phlebotomy Study of Testosterone Undecanoate
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clarus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CLAR-15013
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Results first posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — testosterone undecanoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral Testosterone Undecanoate (Experimental): A single dose of oral testosterone undecanoate equivalent to 200 mg of testosterone in the form of two soft gelatin capsules containing 158 mg of testosterone undecanoate will be administered to each subject.
  Interventions: Drug: Oral Testosterone Undecanoate

INTERVENTIONS:
Drug: Oral Testosterone Undecanoate — Subjects will receive a single dose containing 158 mg of testosterone undecanoate, equivalent to 200 mg testosterone.
  Other Names: testosterone undecanoate

SUMMARY:
An open-label, single oral TU dose study was conducted in eight (8) hypogonadal men at a single study site. Each study participant received a single oral TU dose immediately prior to a standardized breakfast meal comprised of 800 to 1000 calories and approximately 30 g of fat. Blood samples were collected 30 minutes prior dose administration and at 0 pre-dose and post dose at the following hours post-dose; 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours.

DETAILED DESCRIPTION:
This open-label, single oral dose, phlebotomy study was designed to clarify the issue of the influence of blood collection tubes on T, DHT, TU and DHTU measurements by collecting blood samples into various collection tubes from a small number of hypogonadal men dosed with a single oral TU dose in the form of a SEDDS formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Male, 18 to 65 years of age, inclusive, with a diagnosis of hypogonadism and a screening total serum T of < 300 ng/dL.
2. Adequate venous access to allow blood sample collections via venous cannula.
3. Naïve to androgen-replacement therapy or willing to temporarily cease current T treatment and willing to remain off all forms of T except for study medication throughout study.
4. Voluntarily provide written informed consent to participate in this study.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria will not be eligible:

1. Significant intercurrent disease (especially liver, kidney, heart disease, uncontrolled diabetes mellitus or psychiatric illness)
2. Abnormal prostate digital rectal examination, elevated PSA (PSA > 4 ng/mL), AUA Symptom Score ≥ 15 points and/or history of prostate CA.
3. BMI less than 18 kg/m2 or greater than 37 kg/m2
4. Serum transaminases > 2 times upper limit of normal (ULN) or serum bilirubin >2.0 mg/dL.
5. History of severe or multiple allergies, or severe adverse drug reaction. A known hypersensitivity to lidocaine or all surgical dressings which may be used in the study procedures.
6. History of abnormal bleeding tendencies or thrombophlebitis unrelated to venipuncture or intravenous cannulation.
7. Oral, topical or buccal T therapy within previous one week, or intramuscular T injection within previous 4 weeks.
8. Parenteral T-undecanoate therapy within the past 6 months.
9. Use of dietary supplements that may increase serum T, within previous 4 weeks.
10. Known malabsorption syndrome and/or current treatment with oral lipase inhibitors, bile acid-binding resins, colestipol, fibric acid derivatives, clofibrate, gemfibrozil, and probucol.
11. Smokers unable to refrain from smoking during required confinement period.
12. History of, or current evidence of, abuse of alcohol or any drug substance.
13. Receipt of any research study drug within 30 days of study.
14. Blood donation within the 12 week period before the initial study dose.
15. Hematocrit less than 35% or greater than 50%.
16. History of clinically significant polycythemia following treatment with a testosterone replacement product.
17. Current use of paroxetine, clomipramine, antiandrogens, estrogens, potent P450 enzyme inducers, or barbiturates.
18. History of uncontrolled sleep apnea.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Wang, M.D., Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Los Angeles Biomedical Research Institute, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be provided to each respective investigator at the end of the trial.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Testosterone Undecanoate
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oral Testosterone Undecanoate
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: % of Mean Difference in T Concentration Compared to Plain Collection Tube
Description: The measured outcome presented is the difference as a percent of mean of T results when comparing T Concentrations measured in three different types of NaF containing collection tubes (NaF+EDTA, NaF+Oxalate and NaF) to T measured in blood collected in plain tubes. The % of Mean Difference in T concentration for each tube type was obtained by taking the average at each time point a T concentration was obtained, and calculating the mean difference between the test ((NaF+EDTA, NaF+Oxalate and NaF) tubes and the control (plain) tube.
  The concentration of total T will be determined in the serum/plasma samples of all subjects using validated LC/MS/MS methods at the Endocrine and Metabolic Research Lab.
Time Frame: Sample collection at -0.5, and 0 hours pre-dose and post-dose samples collected at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12, hours after a single dose of oral TU.
Measure: Mean (Standard Deviation); unit: Difference as % of Mean of T results
Arm/Group | Oral Testosterone Undecanoate
Number analyzed (Participants) | 8
Difference as % of Mean of T results
  NAF+EDTA | 8.6 (18.3)
  NAF+Oxalate | 16.6 (18.5)
  NAF | 23.2 (20.9)

ADVERSE EVENTS:
Time Frame: 2 months
Description: All adverse events whether causally related to treatment or not are recorded beginning with date of information consent (prior to treatment) and for 7 days following last dose of study drug. Observation period lasted 2 months
Arm/Group | Oral Testosterone Undecanoate
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes